CLINICAL TRIAL: NCT00836082
Title: A Phase 1, Double-Blind (Sponsor Open), Randomised, Placebo-Controlled, Parallel Group, Oral Multiple-Dose Trial To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-04457845 In Healthy Volunteers
Brief Title: A Multiple Dose Trial Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-04457845 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B0541002
Record Dates: First submitted 2009-01-12; First posted 2009-02-04 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Acute Pain; Chronic Pain
Keywords: Healthy volunteers
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (N=10) (Experimental): Placebo-controlled, escalating multiple doses of 0.5mg per day for 14 days.
  Interventions: Drug: PF-04457845, FAAH inhibitor
- Cohort 2 (N=10) (Experimental): Placebo-controlled, escalating multiple doses of 1mg per day for 14 days.
  Interventions: Drug: PF-04457845, FAAH inhibitor
- Cohort 3 (N=10) (Experimental): Placebo-controlled, escalating multiple doses of 4mg per day for 14 days.
  Interventions: Drug: PF-04457845, FAAH inhibitor
- Cohort 4 (N=10) (Experimental): Placebo-controlled, escalating multiple doses of 8mg per day for 14 days.
  Interventions: Drug: PF-04457845, FAAH inhibitor

INTERVENTIONS:
Drug: PF-04457845, FAAH inhibitor — Oral solution of 0.5mg given once daily for 14 days.
  Arms: Cohort 1 (N=10)
Drug: PF-04457845, FAAH inhibitor — Oral solution of 1mg given once daily for 14 days.
  Arms: Cohort 2 (N=10)
Drug: PF-04457845, FAAH inhibitor — Oral solution of 4mg will be administered as a single dose 7-14 days prior to the multiple dosing phase where 4mg will be administered once daily for 14 days.
  Arms: Cohort 3 (N=10)
Drug: PF-04457845, FAAH inhibitor — A randomized food treatment will be administered 7-14 days prior to and on day 1 of the multiple dosing phase
  Arms: Cohort 3 (N=10)
Drug: PF-04457845, FAAH inhibitor — Oral solution of 8mg will be administered as a single dose 7-14 days prior to the multiple dosing phase where 8mg will be administered once daily for 14 days.
  Arms: Cohort 4 (N=10)
Drug: PF-04457845, FAAH inhibitor — A randomized food treatment will be administered 7-14 days prior to and on day 1 of the multiple dosing phase
  Arms: Cohort 4 (N=10)

SUMMARY:
To determine if PF-04457845 at doses of 0.5mg, 1mg, 4mg, and 8 mg given once daily for 14 days will be safe and well tolerated in healthy volunteers. To determine the effect on food on PF-04457845 pharmacokinetics and safety following administration of single doses of 4mg and 8mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects (of non childbearing potential) between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including hyperlipidemia), pancreatic, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* History of febrile illness within 5 days prior to the first dose.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 30 days ( or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec at screening. If QTc exceeds 450msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Females of childbearing potential.
* Use of prescription or nonprescription drugs, and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements and hormonal replacement therapy must be discontinued 28 days prior to the first dose of study medication. As an exception, ibuprofen may be used at doses of up to 1800 mg/day with food. Limited use of non-prescription medications that are not believed to affect subject safety or overall results of the study may be permitted on a case -by-case basis following approval by the sponsor.
* Unwillingness to refrain from consumption of grapefruit or grapefruit/pomelo containing products within 7 days prior to the first dose of study medication until the completion of the follow-up visit.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Subject is the Investigator or sub-Investigator. research assistant, pharmacist, study coordinator, other staff, or a relative of study personnel directly involved with the conduct of the study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* The use of marijuana (or other illicit drugs) within 30 days of randomization.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To characterize the multiple-dose pharmacokinetics of PF-04457845. | 14 Days
To characterize the relationship between PF-04457845 and the level of anandamide and level of FAAH enzyme inhibition in healthy adult volunteers following multiple dosing. | 14 Days
To evaluate the safety and tolerability of multiple oral doses of PF-04457845. | 14 Days
To determine the effect on food on PF-04457845 pharmacokinetics following administration of single doses of 4mg and 8mg. | 7-14 Days
To determine the effect on food on PF-04457845 safety following administration of single doses of 4mg and 8mg. | 7-14 Days

SECONDARY OUTCOMES:
CogState/GMLT | 14 Days
Telemetry | 14 Days
Neurologic Exam | 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0541002&StudyName=A%20multiple%20dose%20trial%20evaluating%20the%20safety%2C%20tolerability%2C%20pharmacokinetics%20and%20pharmacodynamics%20of%20PF-04457845%20in%20healthy%20volunteers